CLINICAL TRIAL: NCT03070483
Title: Blood Pressure in Blacks and Calcium (BBC) and Vitamin D Study
Acronym: BBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Holly J. Mattix-Kramer, Associate Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 209476
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-04

CONDITIONS: Hypertension; Vitamin D Deficiency
MeSH Terms: conditions — Hypertension; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This pilot study is a one arm study which will assess the safety and feasibility of supplementing 15 young adults with African ancestry and low vitamin D levels with 5,000 IU of Cholecalciferol (vitamin D3) combined with 1000 mg of elemental calcium daily for 3 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vitamin D (Experimental): Participants will all receive supplementation with cholecalciferol 5000 IU and calcium citrate 1000 mg daily for 3 months
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 5000 IU cholecalciferol with 1000 mg calcium citrate daily
  Other Names: Vitamin D3

SUMMARY:
Adequate levels of vitamin D are essential for bone health at all ages but low levels of vitamin D may also negatively impact other aspects of health such as blood pressure. The investigators have previously shown that adults with African ancestry living near the equator have much higher levels of vitamin D and higher levels of blood pressure compared to adults with African ancestry living in the Chicago area. Multiple clinical trials have examined vitamin D supplementation for reducing blood pressure levels but very few studies have focused on adults with African ancestry and low vitamin D levels. In addition, most previous clinical trials have not addressed calcium intake. While vitamin D may modulate blood pressure via its actions on activation of the renin angiotensin aldosterone system, it is also possible that vitamin D mediates blood pressure via its effects on gastrointestinal calcium absorption. This pilot study is a one arm study, which will assess the safety and feasibility of supplementing 15 young adults with African ancestry and low vitamin D levels with 5,000 IU of Cholecalciferol (vitamin D3) combined with 1000 mg of elemental calcium daily for 3 months. Participants will be recruited from the Maywood Illinois and surrounding areas with flyers and brochures. The investigators will also contact previous participants of the Modeling the Epidemiologic Study/Vitamin D Ancillary Study by phone and letters. At baseline, all participants will have blood pressure measured and will provide a fasting serum specimen and a 24-hour urine collection. Calcium, parathyroid hormone level vitamin D will be measured in serum specimens and 24-hour urine calcium excretion will be measured. Repeat visits will be completed at 6 and 12 weeks of follow-up to again measure resting blood pressure and serum calcium and vitamin D levels. The overall goal is to collect pilot data to help design a larger trial of vitamin D and calcium supplementation for lowering blood pressure in young adults with African ancestry.

DETAILED DESCRIPTION:
This pilot study will recruit 15 black U.S. adults ages 25-45 years of age with 25(OH)D levels < 20 ng/ml and no use of anti-hypertensive medications and a resting seated systolic blood pressure ≥ 120 mmHg and will measure baseline levels of total 25(OH)D, 25(OH)D2, 25(OH)D3, free vitamin 25(OH)D, active vitamin D [1,25(OH)D], parathyroid hormone level, serum calcium, and 24-hour calcium excretion.

Participants will then take the supplements vitamin D3 5000 IU and elemental calcium 1000 mg daily for three months. Investigators will measure changes in blood pressure, total 25(OH)D, 25(OH)D2 and 25(OH)D3, 1,25(OH)D and free 25(OH)D, parathyroid hormone levels, serum calcium and 24-hour urine calcium excretion over the three month period.

The overall goal is to collect pilot data to determine the feasibility of a larger trial to determine whether vitamin D combined with calcium lowers blood pressure in young black adults with low 25(OH)D levels.

This will be a single arm non-blinded feasibility study of 15 participants. The study population will consist of 15 adults ages 25-45 years with self-reported African American race/ethnicity. All participants will provide written informed consent.

Intervention:

This study has only one arm and all participants will receive Cholecalciferol (vitamin D3) 5,000 IU daily for 3 months and 1000 mg of calcium citrate daily for 3 months. There will be no placebo and no blinding of the agent. Participants will receive a 3 month supply of drugs which will be administered by the Loyola pharmacy. Serum vitamin D and calcium levels will be measured at study initiation and at 6 and 12 weeks (study end). Participants will stop taking stop both vitamin D and calcium administration with serum calcium levels are greater than or equal to 10.6 meq/L and/or a 25(OH)D levels are greater than or equal to 80 ng/dl at the 6 week visit.

Safety Monitoring:

The investigators will query any hospitalizations or emergency room visits over the past month and reasons for those visits at the baseline, 6 and 12 week follow-up visits. Serum calcium and vitamin D levels will be measured at 6 and 12 weeks and anyone with serum calcium levels ≥ 10.6 meq/L and/or a 25(OH)D level ≥ 80 ng/ml will stop treatment. All adverse events will be reported to the Loyola University Chicago Health Sciences Institutional Review Board. A data safety and monitoring board will review all data collected after completion of the 6 week visit to ensure safety of the study.

Stopping plans:

Any participant who develops a serum calcium levels ≥ 10.6 meq/L and/or a 25(OH)D level ≥ 80 ng/ml will stop treatment but they will continue to be monitored in the study through week 12 when serum calcium and 25(OH)D levels will be measured at the end of the study. The study will continue until participants have been followed for 12 weeks.

Analysis Plan:

This feasibility study will examine multiple aspects of the pilot data including the total number of persons enrolled vs. number of total persons identified as eligible. Pill counts will be done at the 6 and 12 week visit to assess compliance with vitamin D and calcium supplementation. The percentage of participants taking 80% or more of the vitamin D3 supplement and the calcium supplement will be determined. The number of participants reporting symptoms and all adverse events will be quantified. Repeated measures analysis of variance models will be used to assess change in the outcome measures including systolic and diastolic blood pressure, vitamin D measures, parathyroid hormone levels and 24-hour urine calcium excretion values.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-45 years
2. Self-reported race/ethnicity African American
3. BMI ≥ 18 kg/m2
4. Total 25(OH)D levels < 20 ng/ml (50 nmol/L)
5. No use of vitamin D supplements within past 30 days of the screening visit
6. Able to provide written informed consent
7. Willing to take a vitamin D supplement daily for 3 months
8. Willing to return for follow-up visits to measure blood pressure and provide a blood sample to measure vitamin D and serum calcium
9. No current use of blood pressure lowering medications
10. Systolic blood pressure ≥ 100 mmHg and diastolic blood pressure ≥ 60 mmHg

Exclusion Criteria:

1. Medical history of chronic disease that affect gastrointestinal absorption of vitamin D: Crohn's disease, cystic fibrosis, and celiac disease
2. Use of medications which may affect total 25(OH)D levels: antiepileptic drugs, steroids, bile acid sequestrants, lipase inhibitors, orlistat
3. Current use of vitamin D supplements or use in past month and unwillingness to discontinue for at least 1 month prior to study enrollment
4. History of kidney stones or hypercalciuria
5. Fasting serum calcium ≥ 10.2 mg/dl
6. Average systolic blood pressure ≥ 140 mmHg
7. Average diastolic blood pressure ≥ 90 mmHg
8. Presence of type 1 diabetes mellitus, active malignancy, active thyroid disease or sarcoidosis
9. Pregnant or planning a pregnancy
10. Estimated glomerular filtration rate (based on serum creatinine level) is < 60 ml/min/1.73 m2 based on the Modification of Diet in Renal Disease formula

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Kramer, MD MPH, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiang D, Kramer H, Luke A, Cooper R, Aloia J, Bovet P, Plange-Rhule J, Forrester T, Lambert V, Camacho P, Dugas L, Durazo-Arvizu R. 25-Hydroxyvitamin D and blood pressure: a plateau effect in adults with African ancestry living at different latitudes. J Hypertens. 2017 May;35(5):968-974. doi: 10.1097/HJH.0000000000001263. PMID 28118279

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D Arm: All participants received cholecalciferol 5000 IU orally and calcium citrate 1000 mg orally daily for 12 weeks
Period: Overall Study
Arm/Group | Vitamin D Arm
Started (First person was screened March 25, 2018) | 5
Completed (Completed the trial) | 3
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 38.4 [27 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Mean arterial blood pressure [Mean (Full Range); unit: mmHg] | 90 [80 to 104]

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Blood Pressure From Baseline to 12 Weeks
Description: Seated blood pressure is measured at baseline and at 6 and 12 week follow-up visits in the clinic using an appropriate sized cuff after a rest period using an automated device (Omron). Blood pressure will be measured three times in one minute intervals at each time point and the average of these three recordings will be recorded as the mean blood pressure at each time point. Arm circumference will be measured to ensure the correct cuff size is used for all blood pressure measurements including home monitoring of blood pressure. Due to small number of participants, the change in mean blood pressure was analyzed as difference in mean blood pressure (2 x average diastolic blood pressure + average systolic blood pressure)/3 between baseline and at 12 weeks.
Time Frame: Difference in BP from baseline and 12 weeks after initiation of intervention
Measure: Mean (Full Range); unit: mmHg
Groups:
- Vitamin D Arm: All participants received vitamin D and calcium supplementation
Arm/Group | Vitamin D Arm
Number analyzed (Participants) | 3
mmHg | 4.3 [2 to 10]

2. Secondary Outcome: Change in Total 25-hydroxyvitamin D From Baseline to 12 Weeks
Description: Total 25-hydroxyvitamin D will be measured with the use of liquid chromatography-tandem mass spectrometry
Time Frame: Change in total 25-hydroxyvitamin D level from baseline to 12 weeks after initiation of intervention
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Vitamin D Arm
Number analyzed (Participants) | 3
ng/ml | 21.7 [9 to 39]

3. Secondary Outcome: Change in Free 25-hydroxyvitamin D Levels From Baseline to 12 Weeks
Description: Free 25(OH)D levels-will be measured using kits from Future Diagnostics (Wijchen, The Netherlands).
Time Frame: Baseline and at 12 weeks after initiation of intervention
Population: We did not measure free vitamin D and only measured total vitamin D because we ran out of funding
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Intact Parathyroid Hormone Levels From Baseline to 12 Weeks
Description: Intact parathyroid hormone levels will be measured with the use of the Elecsys Parathyroid Hormone Immunoassay
Time Frame: Change in PTH levels from baseline and at 12 weeks after initiation of intervention
Population: 3 participants who completed the trial
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Vitamin D
Number analyzed (Participants) | 3
pg/ml | 27.5 [13.0 to 52.5]

5. Secondary Outcome: Change in 1,25-dihydroxyvitamin D From Baseline to 12 Weeks
Description: 1,25 -dihydroxyvitamin D will be measured with the use of liquid chromatography-tandem mass spectrometry
Time Frame: Change in 1,25 dihydroxyvitamin D levels from baseline and at 12 weeks after initiation of intervention
Population: 1,25 vitamin D was never measured due to lack of funding
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in 24-hour Urine Calcium Excretion From Baseline to 12 Weeks
Description: A 24-hour urine will be collected and calcium will be measured by Quest diagnostics
Time Frame: Change in 24 hour urine calcium excretion from baseline and at 12 weeks after initiation of intervention
Population: 3 participants who completed the trial
Measure: Median (Inter-Quartile Range); unit: mg/day
Arm/Group | Vitamin D
Number analyzed (Participants) | 3
mg/day | 336.2 [-6.0 to 632.6]

ADVERSE EVENTS:
Time Frame: 12 weeks of the trial
Description: Hospitalizations or emergency room visits were queried at the 6 and 12 week follow-up visits. Serum calcium and vitamin D levels were measured at 6 and 12 weeks to assess for hypercalcemia defined as serum calcium level 10.6 mg/dl or higher.
Arm/Group | Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
We only enrolled 5 participants and 3 completed the trial. The early termination led to small number of subjects analyzed. We did not measure free vitamin D or 1,25 vitamin D levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03070483/Prot_SAP_000.pdf